CLINICAL TRIAL: NCT00290342
Title: A Multicentric Study to Compare the Immunogenicity, Safety & Reactogenicity of GSK Biologicals' DTPa-IPV Vaccine vs. Co-administration of GSK's DTPa Vaccine & Sanofi-Pasteurs' IPV Vaccine at Different Injection Sites, to Healthy Children
Brief Title: Evaluation of the Immunogenicity, Safety and Reactogenicity of the Combined DTPa-IPV Vaccine in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 104871
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-02

CONDITIONS: Tetanus; Acellular Pertussis; Diphtheria
MeSH Terms: conditions — Tetanus; Diphtheria | interventions — DTPa-HBV-IPV combined vaccine; Pentetic Acid; Diphtheria-Tetanus-acellular Pertussis Vaccines

ARMS (2):
- Infanrix-IPV Group (Experimental): Healthy male or female subjects between and including 8 to 12 weeks (56-90 days) of age at the time of the first vaccination, who were born after a gestation period of 36 to 42 weeks, received 3 doses of the GSK Biologicals' combined Infanrix™-IPV (DTPa-IPV) vaccine at 2, 4 and 6 months of age, intramuscularly into the antero-lateral thigh.
  Interventions: Biological: DTPa-IPV
- Infanrix + IMOVAX Polio Group (Active Comparator): Healthy male or female subjects between and including 8 to 12 weeks (56-90 days) of age at the time of the first vaccination, who were born after a gestation period of 36 to 42 weeks, received 3 doses of the GSK Biologicals' Infanrix™ (DTPa) vaccine co-administered with Sanofi-Pasteur's IMOVAX Polio® (IPV) vaccine at 2, 4 and 6 months of age, intramuscularly into the antero-lateral sides of opposite thighs.
  Interventions: Biological: DTPa; Biological: IMOVAX Polio®

INTERVENTIONS:
Biological: DTPa-IPV — 3 intramuscular injections
  Other Names: Infanrix™-IPV
  Arms: Infanrix-IPV Group
Biological: DTPa — 3 intramuscular injections
  Other Names: Infanrix™
  Arms: Infanrix + IMOVAX Polio Group
Biological: IMOVAX Polio® — 3 intramuscular injections
  Arms: Infanrix + IMOVAX Polio Group

SUMMARY:
DTPa and IPV vaccines are recommended for immunization of infants in Korea. The use of combination vaccines simplifies routine paediatric vaccination. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Participants in this Phase IIIb study will either receive GSK Biologicals' combined diphtheria-tetanus-acellular pertussis-inactivated poliovirus (DTPa-IPV) vaccine or co-administration of GSK Biologicals' combined diphtheria-tetanus-acellular pertussis (DTPa) vaccine and Sanofi-Pasteurs' inactivated poliovirus vaccine. Vaccines for both groups will be administered at 2, 4 and 6 months of age. Two blood samples will be collected during the course of the study: prior to vaccination and one month after the third vaccine dose.

ELIGIBILITY:
Inclusion criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol .
* A male or female between, and including, 8 and 12 weeks (56-90 days) of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Administration of any vaccine within 30 days (i.e.30 days to 1 day) before the first dose of the study vaccine.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the study period (i.e. Day 0 to Month 7), with the exception of Bacille Calmette-Guérin (BCG) vaccine, hepatitis B vaccine, pneumococcal vaccine, flu vaccine and Hib vaccine.
* Planned administration/ administration of a vaccine foreseen by the study protocol (i.e. BCG vaccine, hepatitis B vaccine, pneumococcal, flu vaccine and Hib vaccine) during the period 30 days before and one week after the study vaccine dose.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Previous vaccination against diphtheria, tetanus, pertussis and/or poliovirus disease.
* History of diphtheria, tetanus, pertussis and/or poliovirus diseases.
* Known exposure to diphtheria, tetanus, pertussis and/or poliovirus before the study period.
* Any anaemia/ thrombocytopenia or blood clot that leads to prohibition from intramuscular injection.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 8 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 458 (Actual)
Dates: Start 2006-01-01; Primary Completion 2007-01-01 (Actual); Study Completion 2007-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- South Korea (6):
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 104871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 104871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104871 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 458 subjects enrolled in the study, 6 subjects (5 from Infanrix-IPV Group and 1 from Infanrix + IMOVAX Polio Group) were not administered the study vaccine due to consent withdrawal from parents/guardians and received an elimination code.
Period: Overall Study
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Started | 224 | 228
Completed | 217 | 223
Not Completed | 7 | 5
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group | Total
Number analyzed (Participants) | 224 | 228 | 452
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.8 (0.9) | 8.8 (0.91) | 8.8 (0.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 110 | 222
  Male | 112 | 118 | 230

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroprotected Subjects Against Diphtheria (Anti-D) and Tetanus (Anti-T)
Description: A seroprotected subject was defined as a vaccinated subject with anti-diphteria (anti-D) and anti-tetanus (anti-T) antibody concentrations greater than or equal to (≥) the cut-off value of 0.1 international units/milliliter (IU//mL).
Time Frame: One month (Month 5) post-primary vaccination course
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 204 | 211
Subjects
  Anti-D | 204 | 211
  Anti-T | 204 | 211
Statistical Analysis 1: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Non-inferiority in terms of vaccine response to diphteria; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to diphtheria, standardized asymptotic 95% CI for the groups'difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-1.85 to 1.79]
Statistical Analysis 2: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Non-inferiority in terms of vaccine response to tetanus; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to tetanus, standardized asymptotic 95% CI for the groups'difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-1.85 to 1.79]

2. Primary Outcome: Number of Seroprotected Subjects Against Poliovirus (Anti-polio) Types 1, 2 and 3
Description: A seroprotected subject was defined as a vaccinated subject with anti-poliovirus types 1, 2 and 3 (Anti-Polio 1, 2 and 3) antibody titers greater than or equal to (≥) the cut-off value of 8.
Time Frame: One month (Month 5) post-primary vaccination course
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 204 | 207
Subjects
  Anti-polio 1 (N=204; 207) | 204 | 207
  Anti-polio 2 (N=204; 205): number analyzed (Participants) | 204 | 205
  Anti-polio 2 (N=204; 205) | 204 | 204
  Anti-polio 3 (N=204; 207) | 203 | 206
Statistical Analysis 1: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Immune response non-inferiority - Anti-Polio 1; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to poliovirus type 1, standardized asymptotic 95% CI for the groups' difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = 0, 95% CI 2-sided [-1.85 to 1.82]
Statistical Analysis 2: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Immune response non-inferiority - Anti-Polio 2; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to poliovirus type 2, standardized asymptotic 95% CI for the groups' difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = 0.49, 95% CI 2-sided [-1.36 to 2.71]
Statistical Analysis 3: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Immune response non-inferiority - Anti-Polio 3; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to poliovirus type 3, standardized asymptotic 95% CI for the groups' difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = -0.01, 95% CI 2-sided [-2.28 to 2.24]

3. Primary Outcome: Number of Subjects With a Vaccine Response for Anti-pertussis Toxoid (Anti-PT), Anti-pertactin (Anti-PRN) and Anti-filamentous Haemagglutinin (Anti-FHA)
Description: Vaccine response was defined as: - for initially seronegative subjects, antibody concentrations ≥ 5 EL.U/mL one month after third vaccine dose; - for initially seropositive subjects, at least maintenance of pre-vaccination antibody concentrations one month after third vaccine dose.
Time Frame: One month (Month 5) post-primary vaccination course
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 202 | 211
Subjects
  Anti-PT: number analyzed (Participants) | 200 | 209
  Anti-PT | 200 | 206
  Anti-FHA | 201 | 209
  Anti-PRN | 202 | 210
Statistical Analysis 1: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Immune response non-inferiority - Anti-PT; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to pertussis toxoid, standardized asymptotic 95% CI for the groups' difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = 1.44, 95% CI 2-sided [-0.46 to 4.13]
Statistical Analysis 2: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Immune response non-inferiority - Anti-FHA; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to filamentous haemagglutinin, standardized asymptotic 95% CI for the groups' difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = 0.45, 95% CI 2-sided [-1.88 to 2.95]
Statistical Analysis 3: Comparison: Infanrix-IPV Group vs Infanrix + IMOVAX Polio Group; Immune response non-inferiority - Anti-PRN; Test type: Non-Inferiority or Equivalence — To assess the non-inferiority of the Infanrix-IPV Group compared to the Infanrix + IMOVAX Polio Group in terms of vaccine response to pertactin, standardized asymptotic 95% CI for the groups' difference (Infanrix-IPV Group minus Infanrix + IMOVAX Polio Group) was computed. Objective of non-inferiority was met since the LL of the 95% CI was above -10%; Difference in seroprotection rate = 0.47, 95% CI 2-sided [-1.4 to 2.64]

4. Primary Outcome: Number of Subjects With Vaccine Response to Pertussis Toxoid (PT), Pertactin (PRN) and Filamentous Haemagglutinin (FHA) Antigens
Description: Vaccine response to pertussis toxoid (PT), pertactin (PRN) and filamentous haemagglutinin (FHA) was defined as the appearance of antibodies in subjects who were initially (i.e. before vaccination) seronegative (i.e. with concentrations < 5 EL.U/mL), or at least as the maintenance of pre-vaccination antibody concentrations in subjects who were initially seropositive (i.e. with concentrations ≥ 5 EL.U/mL value).
Time Frame: One month (Month 5) post-primary vaccination course
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 202 | 211
Subjects
  Anti-PT (N=200; 209): number analyzed (Participants) | 202 | 209
  Anti-PT (N=200; 209) | 200 | 206
  Anti-FHA (N=202; 211) | 201 | 209
  Anti-PRN (N=202; 211) | 202 | 210

5. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria (Anti-D) and Tetanus (Anti-T)
Description: A seroprotected subject was defined as a vaccinated subject with anti-diphteria (anti-D) and anti-tetanus (anti-T) antibody concentrations greater than or equal to (≥) the cut-off value of 1 international units/milliliter (IU//mL).
Time Frame: Before (Pre) and one month after (Post) the primary vaccination course
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 204 | 212
Subjects
  Anti-D, PRE (N=202; 212): number analyzed (Participants) | 202 | 212
  Anti-D, PRE (N=202; 212) | 0 | 0
  Anti-D, POST (N=204; 211): number analyzed (Participants) | 204 | 211
  Anti-D, POST (N=204; 211) | 194 | 187
  Anti-T, PRE (N=202; 212): number analyzed (Participants) | 202 | 212
  Anti-T, PRE (N=202; 212) | 1 | 1
  Anti-T, POST (N=204; 211): number analyzed (Participants) | 204 | 211
  Anti-T, POST (N=204; 211) | 204 | 208

6. Secondary Outcome: Concentration of Antibodies Against Diphteria (Anti-D) and Tetanus (Anti-T)
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in international units per millilitre (mIU/mL).
Time Frame: Before (Pre) and one month after (Post) the primary vaccination course
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 204 | 212
IU/mL
  Anti-D, PRE (N=202; 212): number analyzed (Participants) | 202 | 212
  Anti-D, PRE (N=202; 212) | 0.052 [0.051 to 0.054] | 0.053 [0.05 to 0.055]
  Anti-D, POST (N=204; 211): number analyzed (Participants) | 204 | 211
  Anti-D, POST (N=204; 211) | 4.333 [3.902 to 4.813] | 2.63 [2.36 to 2.932]
  Anti-T, PRE (N=202; 212): number analyzed (Participants) | 202 | 212
  Anti-T, PRE (N=202; 212) | 0.059 [0.055 to 0.064] | 0.06 [0.056 to 0.065]
  Anti-T, POST (N=204; 211): number analyzed (Participants) | 204 | 211
  Anti-T, POST (N=204; 211) | 10.306 [9.5 to 11.18] | 7.139 [6.512 to 7.826]

7. Secondary Outcome: Titers for Poliovirus Type 1, 2 and 3 Antibodies
Description: Titers for anti-polio 1, 2 and 3 are presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was greater than or equal to (≥) 8.
Time Frame: Before (Pre) and one month after (Post) the primary vaccination course
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 204 | 212
Titers
  Anti-polio 1, PRE (N=199; 212): number analyzed (Participants) | 199 | 212
  Anti-polio 1, PRE (N=199; 212) | 6.3 [5.5 to 7.1] | 6.1 [5.4 to 6.9]
  Anti-polio 1, POST (N=204; 207): number analyzed (Participants) | 204 | 207
  Anti-polio 1, POST (N=204; 207) | 755.7 [643.5 to 887.4] | 263 [232.1 to 298]
  Anti-polio 2, PRE (N=202; 211): number analyzed (Participants) | 202 | 211
  Anti-polio 2, PRE (N=202; 211) | 5.8 [5.2 to 6.5] | 6.5 [5.8 to 7.3]
  Anti-polio 2, POST (N=204; 205): number analyzed (Participants) | 204 | 205
  Anti-polio 2, POST (N=204; 205) | 704.7 [599.5 to 828.4] | 267.6 [233.4 to 306.8]
  Anti-polio 3, PRE (N=202; 212): number analyzed (Participants) | 202 | 212
  Anti-polio 3, PRE (N=202; 212) | 5 [4.5 to 5.4] | 4.9 [4.5 to 5.3]
  Anti-polio 3, POST (N=204; 207): number analyzed (Participants) | 204 | 207
  Anti-polio 3, POST (N=204; 207) | 1209.5 [1040.1 to 1406.5] | 438.3 [383.1 to 501.3]

8. Secondary Outcome: Concentrations of Antibodies Against Pertussis Toxoid (Anti-PT), Pertactin (Anti-PRN) and Filamentous Haemagglutinin (Anti-FHA)
Description: Concentrations are presented as geometric mean concentrations (GMCs), expressed in ELISA units per millilitre (EL.U/mL).
Time Frame: Before (Pre) and one month after (Post) the primary vaccination course
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 204 | 212
EL.U/mL
  Anti-PT, PRE (N=200; 210): number analyzed (Participants) | 200 | 210
  Anti-PT, PRE (N=200; 210) | 3 [2.8 to 3.2] | 3.2 [3 to 3.5]
  Anti-PT, POST (N=204; 211): number analyzed (Participants) | 204 | 211
  Anti-PT, POST (N=204; 211) | 63.3 [58.7 to 68.2] | 55.6 [50.9 to 60.7]
  Anti-FHA, PRE (N=202; 212): number analyzed (Participants) | 202 | 212
  Anti-FHA, PRE (N=202; 212) | 7.4 [6.5 to 8.4] | 8.5 [7.4 to 9.7]
  Anti-FHA, POST (N=204; 211): number analyzed (Participants) | 204 | 211
  Anti-FHA, POST (N=204; 211) | 294.3 [269.5 to 321.4] | 259.6 [235.1 to 286.6]
  Anti-PRN, PRE (N=202; 212): number analyzed (Participants) | 202 | 212
  Anti-PRN, PRE (N=202; 212) | 2.7 [2.5 to 2.8] | 2.7 [2.6 to 2.9]
  Anti-PRN, POST (N=204; 211): number analyzed (Participants) | 204 | 211
  Anti-PRN, POST (N=204; 211) | 205 [187.7 to 223.9] | 155.6 [140.7 to 172.1]

9. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = crying when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: During the 4-day (Days 0-3) post-vaccination period, across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had the symptom sheet filled-in.
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 220 | 226
Subjects
  Any Pain | 92 | 96
  Grade 3 Pain | 5 | 8
  Any Redness | 115 | 116
  Grade 3 Redness | 22 | 26
  Any Swelling | 74 | 79
  Grade 3 Swelling | 17 | 20

10. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 drowsiness = drowsiness that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Grade 3 irritability = crying that could not be comforted/ prevented normal activity. Grade 3 Loss of appetite = not eating at all. Related = symptom symptoms considered by the investigator to have a causal relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period, across doses
Population: as for outcome 9
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 221 | 226
Subjects
  Any Drowsiness | 95 | 99
  Grade 3 Drowsiness | 4 | 2
  Related Drowsiness | 54 | 53
  Any Fever (axillary) | 63 | 38
  Grade 3 Fever (axillary) | 4 | 1
  Related Fever (axillary) | 45 | 22
  Any Irritability | 140 | 139
  Grade Irritability | 14 | 10
  Related Irritability | 85 | 91
  Any Loss of appetite | 84 | 78
  Grade 3 Loss of appetite | 1 | 0
  Related Loss of appetite | 50 | 46

11. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 224 | 228
Subjects | 135 | 138

12. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (from Month 0 up to Month 5)
Population: as for outcome 11
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Number analyzed (Participants) | 224 | 228
Subjects | 15 | 17

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms during the 4-day (Days 0-3) post-vaccination period; Unsolicited AEs during the 31-day (Days 0-30) post-vaccination period and SAEs during the entire study period (from Month 0 up to Month 5)
Arm/Group | Infanrix-IPV Group | Infanrix + IMOVAX Polio Group
Serious Adverse Events (participants affected / at risk) | 15/224 | 17/228
Other Adverse Events (participants affected / at risk) | 200/224 | 196/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV Group (N=224) | Infanrix + IMOVAX Polio Group (N=228)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 1
Febrile convulsion (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 7 | 3
Pneumonia (Infections and infestations) | 4 | 5
Urinary tract infection (Infections and infestations) | 3 | 5
Gastroenteritis (Infections and infestations) | 2 | 2
Kawasaki's disease (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infanrix-IPV Group (N=224) | Infanrix + IMOVAX Polio Group (N=228)
Bronchiolitis (Infections and infestations) | 14 (14) | 7 (11)
Bronchitis (Infections and infestations) | 7 (8) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 84 (130) | 78 (115)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 16 (18) | 17 (20)
Diarrhoea (Gastrointestinal disorders) | 12 (16) | 8 (8)
Erythema (Skin and subcutaneous tissue disorders) | 115 (212) | 116 (209)
Gastroenteritis (Infections and infestations) | 10 (11) | 13 (14)
Irritability (Psychiatric disorders) | 140 (238) | 139 (241)
Pain (General disorders) | 92 (164) | 96 (161)
Pyrexia (General disorders) | 74 (91) | 40 (48)
Somnolence (Nervous system disorders) | 95 (152) | 99 (161)
Swelling (General disorders) | 74 (114) | 79 (129)
Upper respiratory tract infection (Infections and infestations) | 72 (98) | 61 (88)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.